CLINICAL TRIAL: NCT02790801
Title: The First Russian Observational Survey of Heart Failure Patients With Atrial Fibrillation
Acronym: RIF-CHF
Status: Completed | Type: Observational
Sponsor: Federal State Budgetary Scientific Institution, Research Institute of Cardiology (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Sergey Tereschenko, MD,Phd,prof, Head of department, Federal State Budgetary Scientific Institution, Research Institute of Cardiology
Other Study IDs: RW52.1
Record Dates: First submitted 2016-05-31; First posted 2016-06-06 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Chronic Heart Failure; Atrial Fibrillation
Keywords: chronic heart failure; atrial fibrillation; anticoagulant
MeSH Terms: conditions — Atrial Fibrillation | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1 group: observation of patients with chronic heart failure and atrial fibrillation
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — observation

SUMMARY:
The purpose of this study is to evaluate the management of chronic heart failure patients with atrial fibrillation, to collect data on compliance with clinical guidelines and the prevalence of long-term anticoagulant therapy,complications. The results will be used to develop most rational therapeutic and diagnostic strategies to improve clinical outcomes of such patients.

DETAILED DESCRIPTION:
Quality assurance plan: investigators are going to plan site monitoring every three months. Any audits are not planned Investigatirs will check all entered data into the registry with the predefined ranges. The database is protected against any inconsistency and incorrect entering by the strictly predefined range in all fields. Instead of that, data checks will be performed yearly.

During the site monitoring data verification of the transfer from source documents to the database will be performed.

Iiverstigators have data dictionary, which includes descriptions of each variable and, if relevant, normal ranges.

Investigators use standard local operation procedures for any activities during the registry (as patient recruitment, data collection and management, data analysis) and local authorities approve all of those procedures.

Investigators calculated the sample size for demonstration of hypothesis of the registry.

Descriptive analysis of the data will be reported using basic summary statistics. Results will be summarized for the whole group and for the diagnostic subgroups. P-values and confidence intervals will be 2-sided, and statistical significance will be declared at the 2-sided 0,05-level. For continuous variables mean values, standard deviations, 95% confidence intervals, median and lower and upper percentiles, as well as minimum and maximum values will be calculated.

Safety is assessed by reports of AEs with relation, seriousness, action taken, and outcome. AEs are summarized using the MedDRA coding system. Event rates for single AEs are calculated based on the total number of documented patients. AEs are categorized according to relation, seriousness and outcome.

ELIGIBILITY:
Inclusion Criteria:

* patient has symptomatic chronic heart failure diagnosed more than 3 months before enrolling, if ejection fraction of left ventricular is >40% - N terminal-pro-B-type natriuretic peptide should be ≥300 pg/ml or B-type natriuretic peptide ≥100 pg/ml.
* patient has non-valvular stable atrial fibrillation

Exclusion Criteria:

* transient ischemic attack within 3 days before inclusion,
* stroke during 14 days before inclusion,
* myocardial infarction within 14 days before inclusion,
* thromboembolic complications or thrombosis within 14 days before inclusion,
* heart failure because of valvular pathology,
* heart failure induced by infection agents or infiltrative diseases, alcohol consumption, use of psychoactive drugs; peripartal heart failure; transient conditions
* planning heart transplantation
* implantation of biventricular pacemaker within 28 days before inclusion
* any severe condition limiting life less than 3 months
* HIV infection
* Alcohol consumption or psychoactive drugs intake
* participation in any experimental study within 30 days before inclusion
* patient is not ready to contact by telephone at the end of the study at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients from primary care clinics, hospilals
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2015-02; Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with hospitalization for worsening of heart failure. HF hospitalization is defined as an overnight stay, or longer, in a hospital environment due to HF as the primary reason | Day 1 up to approximately 12 months

SECONDARY OUTCOMES:
Death due to a cardiovascular cause. CV mortality is defined as death due to heart failure, myocardial infarction, cardiac arrhythmia, stroke or cerebral vascular accident (CVA), other CV. | Day 1 up to approximately 12 months
All-cause mortality. Death due to any cause. | 1 year
Rate of thromboembolic events defined as ischemic stroke, system embolism, deep vein thrombosis, pulmonary embolism. | Day 1 up to approximately 12 months
Bleeding rate. ISTH major or CRNM bleeding during the time the patient is taking the medicine which is 6 months | 1 year
  Day 1 up to approximately 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sergey N Tereshchenko, Prof, Principal Investigator — Federal State Budgetary Scientific Institution, Research Institute of Cardiology
Locations (1):
- FSSICardiology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] S.N. Tereshchenko, I.V. Zhirov, N.V. Romanova, Yu.F. Osmolovskaya, S.P. Golitsyn. The first Russian register of patients with chronic heart failure and atrial fibrillation (RIF-CHF): study design.Pharmacother Cardiol 2015;11(6):577-581.